CLINICAL TRIAL: NCT05916066
Title: Nicotinamide and Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NAMG2021
Record Dates: First submitted 2021-10-04; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Niacinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy controls (Other): Healthy controls
  Interventions: Dietary Supplement: Nicotinamide
- Pseudoexfoliative glaucoma (Other): PEXG
  Interventions: Dietary Supplement: Nicotinamide
- POAG (Other): POAG
  Interventions: Dietary Supplement: Nicotinamide
- NTG (Other): NTG
  Interventions: Dietary Supplement: Nicotinamide

INTERVENTIONS:
Dietary Supplement: Nicotinamide — Tabletts of 500mg Nicotinamide (B3-vitamin)

SUMMARY:
The investigators will include different subgroups of open-angle glaucoma and healthy controls. The participants will attend two visits with two weeks apart. At each visit the participants will have blood drawn and will undergo OCT examination. In between the two visits, participants will receive a treatment of Nicotinamide 1,5g/day for one week and 3.0g/day for the second week.

DETAILED DESCRIPTION:
The investigators plan to recruit four groups, each containing 30 subjects: 1) pseudoexfoliative glaucoma, 2) High tension open-angle glaucoma, 3) Normal tension glaucoma 4) Age-matched controls. Those enrolled will undergo two visits including an ophthalmic exam, blood sampling, and at the first visit, distribution of nicotinamide tablets. We plan to recruit participants amongst glaucoma patients already followed at the Eye Clinic at Umeå University Hospital. Furthermore, age-matched controls will be recruited through lists from the population register at Statistics Sweden. Before enrolling any subject, they will receive both oral and written information as well as sign a consent form. Furthermore, they will be evaluated to make sure that they fulfill the inclusion- and exclusion criteria prior to inclusion.

The ophthalmic exam includes measurement of IOP, perimetry, and OCT/A. Between visits, the participants will receive 1,5 grams of NAM per day the first week and 3 grams per day the second week. The blood drawn will initially be sent to Biobanken Norr for storage. Samples will then be sent to the Swedish Metabolomics Centre, Umeå University and Department of Medical Biochemistry and Biophysics, Karolinska University for analysis using high-resolution mass spectrometry.

ELIGIBILITY:
Inclusion criteria for glaucoma patients:

* Manifest glaucoma (PEXG, HTG, NTG) in one or two eyes,
* age > 18 years,
* replicable visual field defects that cannot be explained by any other disease or insult,
* suspect/anomalous optic nerve head or abnormalities in the retinal nerve fiber layer.

Inclusion criteria for age-matched controls:

-A normal visual field and optic nerve, age > 18 years.

Exclusion criteria for all:

* Any disease affecting retinal function (such as more than mild macular degeneration or diabetic retinopathy), neurological or other non-glaucomatous conditions that may affect the visual field,
* inability to perform a perimetric exam,
* resistance in quitting intake of multivitamins or B-vitamins,
* allergy to NAM or niacin, previous eye surgery involving the central retina,
* pregnant or breast-feeding women,
* fertile women not using reliable contraception,
* diagnosis of cancer in the last five years (not including treated squamous cell carcinoma), anamnesis of liver-disease or peptic ulcer,
* not able to speak and understand either Swedish or English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-16 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Plasma level of NAM before and after NAM treatment in all groups | Two weeks
  Are NAM levels in plasma lower in patients with glaucoma compared to healthy controls and will a short-term treatment with NAM raise the plasma concentration of NAM?

SECONDARY OUTCOMES:
Perfusion density and flow index in macula and optic nerve head before and after NAM treatment in all gropus | Two weeks
  Will a short-term treatment with NAM influence the retinal vasculature measured with OCTA?

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Science, Ophthalmology, Umeå University, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No